CLINICAL TRIAL: NCT00027027
Title: A Phase I, Open-Label, Multicenter, Dose-Escalation Study of the Safety and Pharmacokinetics of a Recombinant Humanized Antibody to Her2 (rhuMAb 2C4) Administered Every 3 Weeks to Subjects With Advanced Solid Malignancies
Brief Title: Safety Study of rhuMAb 2C4 to Treat Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOC2297g
Record Dates: First submitted 2001-11-15; First posted 2001-11-16 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — pertuzumab

INTERVENTIONS:
Drug: rhuMAb 2C4

SUMMARY:
The purpose of this Phase I study is to test the safety of rhuMAb 2C4 to see what effects (good and bad) it has on patients with certain types of cancer, and also to find the highest dose of rhuMAb that can be given without causing severe side effects. All study participants will be assigned to specific group to evaluate different dosages of rhuMAb 2C4. The study is scheduled to run for up to one year depending on how patients respond to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >=18 years old
* ECOG performance status of 0 or 1 (see Appendix F)
* Life expectancy of >=12 weeks
* Histologically documented, incurable, locally advanced or metastatic solid malignancies
* Disease progression on or after standard effective therapy or a malignancy for which there is no standard therapy
* At least one bi-dimensionally measurable lesion (>=2 cm [>=1 cm on spiral CT scan])
* HER2-negative status as defined by fluorescence in situ hybridization (FISH) testing (only for subjects with breast cancer)
* Use of an effective means of contraception for women of childbearing potential
* Granulocyte count of >=1500/uL, platelet count of >=100,000/uL, and hemoglobin of >=9 g/dL
* Serum bilirubin less than or equal to the upper limit of normal (ULN) and alkaline phosphatase, AST, and ALT <=2.5x ULN (ALT and AST <=5x ULN for subjects with liver metastases; alkaline phosphatase <=5x ULN for subjects with liver or bone metastases)
* Serum creatinine less than or equal to ULN or creatinine clearance of >=60 mL/min
* International normalized ratio (INR) of <1.3 and activated partial thromboplastin time (aPTT) of <1.5x ULN

Exclusion Criteria:

* Pleural effusions, ascites, or bone lesions as the only manifestation of the current cancer
* Symptomatic or untreated brain metastases
* Prior chemotherapy, hormonal therapy (except for androgen-deprivation therapy for subjects with prostate cancer), radiotherapy, or immunotherapy within 4 weeks of Day 1 (within 6 weeks for nitrosoureas or mitomycin)
* Prior treatment with Herceptin
* Prior cumulative doxorubicin dose of >360 mg/m2 or the equivalent
* History of other malignancies within 5 years of Day 1 except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer
* History of significant cardiac disease, unstable angina, congestive heart failure, myocardial infarction, or ventricular arrhythmia requiring medication
* Ejection fraction of <50% or below the lower limit of normal determined by ECHO (Subjects who are unable to have ejection fraction evaluated by ECHO may have ejection fraction evaluated by a MUGA scan, although this must be discussed with the Medical Monitor prior to enrollment.)
* Active infection requiring IV antibiotics
* Uncontrolled hypercalcemia (>11.5 mg/dL)
* Clinically important history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus (HIV) infection
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications
* Major surgery or significant traumatic injury within 3 weeks of Day 1
* Pregnancy or lactation
* Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2001-11; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- rhuMAb 2C4: 0.5 Milligrams Per Kilogram (mg/kg): Recombinant Humanized Antibody to human epidermal growth factor receptor 2 (rhuMAb 2C4) 0.5 mg/kg was administered once every 3 weeks as an intravenous (IV) infusion until progressive disease (PD) or unacceptable toxicity occurred for up to a maximum of 1 year.
- rhuMAb 2C4: 2 mg/kg: rhuMAb 2C4 2 mg/kg was administered once every 3 weeks as an IV infusion until PD or unacceptable toxicity occurred for up to a maximum of 1 year.
- rhuMAb 2C4: 5 mg/kg: rhuMAb 2C4 5 mg/kg was administered once every 3 weeks as an IV infusion until PD or unacceptable toxicity occurred for up to a maximum of 1 year.
- rhuMAb 2C4: 10 mg/kg: rhuMAb 2C4 10 mg/kg was administered once every 3 weeks as an IV infusion until PD or unacceptable toxicity occurred for up to a maximum of 1 year.
- rhuMAb 2C4: 15 mg/kg: rhuMAb 2C4 15 mg/kg was administered once every 3 weeks as an IV infusion until PD or unacceptable toxicity occurred for up to a maximum of 1 year.
Period: Overall Study
Arm/Group | rhuMAb 2C4: 0.5 Milligrams Per Kilogram (mg/kg) | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Started | 3 | 3 | 4 | 3 | 8
Discontinued Before 2 Treatment Cycles | 0 | 0 | 1 | 0 | 1
Completed 2 Cycles of Treatment | 3 | 3 | 3 | 3 | 7
Discontinued at Cycle 2 | 2 | 2 | 1 | 1 | 3
Treated Beyond Cycle 2 | 1 | 1 | 2 | 2 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 3 | 8
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1
Not completed — Admitted for Signs of PD | 0 | 0 | 0 | 0 | 1
Not completed — Clinical Symptoms Progression not PD | 1 | 0 | 0 | 0 | 0
Not completed — PD Requiring Surgery | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision Due To PD | 2 | 3 | 2 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants that were enrolled into one of the 5 treatment groups.
Groups:
- rhuMAb 2C4: 0.5 mg/kg: rhuMAb 2C4 0.5 mg/kg was administered once every 3 weeks as an IV infusion until PD or unacceptable toxicity occurred for up to a maximum of 1 year.
- Total: Total of all reporting groups
Arm/Group | rhuMAb 2C4: 0.5 mg/kg | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (20.4) | 55 (13.6) | 48 (13.8) | 61 (17.1) | 60 (8.2) | 56.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 0 | 6 | 12
  Male | 1 | 2 | 1 | 3 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE), Serious Adverse Event (SAE), or Death
Description: For this protocol, an AE is defined any untoward medical occurrence (e.g., sign, symptom, disease, syndrome, intercurrent illness, abnormal laboratory finding) that emerges or worsens relative to pretreatment baseline during the treatment or post-treatment periods, regardless of the suspected cause.
  For this protocol an SAE was defined as any AE that occurred at any dose if:
  * It resulted in death (i.e., the AE caused or led to death),
  * It was life threatening,
  * It required or prolonged inpatient hospitalization,
  * It was disabling,
  * It resulted in a congenital anomaly/birth defect,
  * It may have jeopardized the participant or may have required medical or surgical intervention to prevent one of the outcomes listed above.
  The primary cause of death for all reported cases was disease progression, and all of the deaths occurred following study discontinuation, with one death occurring within 4 weeks of the last treatment day.
Time Frame: Days 1, 2, 5, 8, and 15 of Cycle 1; Days 1, 8, and Week 3, of Cycles 2 and beyond up to 1 year and at the follow-up visit (4 weeks after last infusion)
Population: All enrolled participants
Measure: Number; unit: participants
Arm/Group | rhuMAb 2C4: 0.5 mg/kg | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 8
participants
  Adverse events | 3 | 3 | 4 | 3 | 8
  Serious adverse events | 3 | 1 | 2 | 0 | 5
  Death | 3 | 1 | 2 | 0 | 1

2. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: Incidence of DLTs defined as any Grade 3 or 4 major organ toxicity according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) Version 2 or any subjectively intolerable toxicity felt by the investigator to be related to rhuMAb 2C4.
  One participant in the 15.0 mg/kg dose group experienced a gastrointestinal hemorrhage on Day 16. This event was judged by the investigator to be related to study drug. The participant recovered in 3 days and continued to receive rhuMAb 2C4 beyond Cycle 2.This was the only DLT reported during the first two treatment cycles.
Time Frame: Day 1 of Cycles 1 and 2, and 24 hours after Cycle 2 infusion
Population: All enrolled participants who completed at least 2 cycles of study treatment.
Measure: Number; unit: participants
Arm/Group | rhuMAb 2C4: 0.5 mg/kg | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 7
participants | 3 | 1 | 2 | 0 | 6

3. Secondary Outcome: Pharmacokinetic Measurement of Area Under the Curve (AUC)
Description: Mean rhuMAb 2C4 serum concentrations versus nominal time profiles for the first two treatment cycles are presented for AUC micrograms per milliliters (ug/mL) by day. A one-compartment model was used for the 0.5 mg/kg dose group, and a two-compartment model was used for the 2-15 mg/kg dose groups.
Time Frame: Days 1 (predose, 89 minutes following start of infusion and at 1.5, 4, and 8 hours postdose) 2, 5, 8 and 15 of Cycle 1; Days 1 (predose and 29 minutes following start of infusion) and 8 of Cycle 2
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: ug*hr/mL
Arm/Group | rhuMAb 2C4: 0.5 mg/kg | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 8
ug*hr/mL | 43.057 (17.770) | 569.433 (168.995) | 1478.000 (349.396) | 3959.333 (1110.113) | 4502.625 (1245.289)

4. Secondary Outcome: Pharmacokinetic Measurement of Systemic Clearance (CL)
Description: A one-compartment model was used for the 0.5 mg/kg dose group, and a two-compartment model was used for the 2-15 mg/kg dose groups.
Time Frame: Days 1 (predose, 89 minutes from infusion start, at 1.5, 4, and 8 hours postdose), 2, 5, 8 and 15 of Cycle 1; Days 1 (predose, 29 minutes from infusion start) and 8 of Cycles 2 and beyond until the follow-up visit (4 weeks after the last infusion)
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | rhuMAb 2C4: 0.5 mg/kg | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 8
mL/day/kg | 13.1 (5.5) | 3.74 (1.28) | 3.52 (0.85) | 2.69 (0.92) | 3.68 (1.47)

5. Secondary Outcome: Pharmacokinetic Measurement of Volume of Central Compartment (Vc)
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | rhuMAb 2C4: 0.5 mg/kg | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 8
mL/kg | 43.6 (4.6) | 35.5 (3.5) | 39.7 (6.2) | 38.4 (5.3) | 42.8 (7.9)

6. Secondary Outcome: Pharmacokinetic Measurement of Steady-State Volume of Distribution (Vss)
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Only participants in the measured treatment groups where a two-compartment model was used are included in the analysis.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 8
mL/kg | 69.5 (13.7) | 74.1 (30.4) | 73.4 (13.6) | 85.3 (36.7)

7. Secondary Outcome: Pharmacokinetic Measurement of Initial Distribution Half-Life (t1/2 Initial)
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Only participants in the measured treatment groups where a two-compartment model was used are included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 8
days | 0.96 (0.99) | 1.09 (0.74) | 1.23 (0.90) | 1.50 (1.17)

8. Secondary Outcome: Pharmacokinetic Measurement of Terminal Half-Life (t1/2 Terminal) in Days
Description: as for outcome 4
Time Frame: as for outcome 4
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: days
Arm/Group | rhuMAb 2C4: 0.5 mg/kg | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 8
days | 2.6 (0.9) | 14.9 (1.1) | 17.2 (10.3) | 22.3 (9.9) | 18.6 (8.8)

ADVERSE EVENTS:
Time Frame: From baseline through 4 weeks after the last infusion of study drug, up to 56 weeks.
Arm/Group | rhuMAb 2C4: 0.5 mg/kg | rhuMAb 2C4: 2 mg/kg | rhuMAb 2C4: 5 mg/kg | rhuMAb 2C4: 10 mg/kg | rhuMAb 2C4: 15 mg/kg
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 2/4 | 0/3 | 5/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rhuMAb 2C4: 0.5 mg/kg (N=3) | rhuMAb 2C4: 2 mg/kg (N=3) | rhuMAb 2C4: 5 mg/kg (N=4) | rhuMAb 2C4: 10 mg/kg (N=3) | rhuMAb 2C4: 15 mg/kg (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rhuMAb 2C4: 0.5 mg/kg (N=3) | rhuMAb 2C4: 2 mg/kg (N=3) | rhuMAb 2C4: 5 mg/kg (N=4) | rhuMAb 2C4: 10 mg/kg (N=3) | rhuMAb 2C4: 15 mg/kg (N=8)
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 1 | 2 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Loose stools (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Anal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral soft tissue disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 1 | 1 | 5
Pyrexia (General disorders) | 2 | 1 | 1 | 0 | 2
Oedema peripheral (General disorders) | 2 | 0 | 0 | 0 | 2
Rigors (General disorders) | 1 | 0 | 1 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0
Gait abnormal (General disorders) | 0 | 0 | 2 | 0 | 0
Malaise (General disorders) | 0 | 0 | 2 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hypotrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Onychorrhexis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Breath sounds decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal passage irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysguesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysgraphia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypoguesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 1 | 2
Alanine aminotranseferase increased (Investigations) | 1 | 0 | 0 | 2 | 1
Aspertate aminotransferase increased (Investigations) | 1 | 1 | 0 | 1 | 1
Troponin T increased (Investigations) | 1 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 0 | 0 | 1
Protein urine (Investigations) | 0 | 1 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Urinary retension (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urethral stricture (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blister (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 0 | 0 | 0 | 0 | 1
Madarosis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Tumor necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Nasal sinus drainage (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.